CLINICAL TRIAL: NCT02575443
Title: Neuromuscular Block and Anesthetic Depth Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Dr, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ADMS NMD depth
Record Dates: First submitted 2015-10-06; First posted 2015-10-14 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Cholecystectomy, Laparoscopic
MeSH Terms: interventions — Rocuronium

ARMS (2):
- Moderate block (MB) group (Experimental)
  Interventions: Drug: Rocuronium (MB group)
- Deep block (DB) group (Experimental)
  Interventions: Drug: Rocuronium (DB group)

INTERVENTIONS:
Drug: Rocuronium (MB group) — Count of train-of-four: 1-2 Titration of rocuronium dose
  Arms: Moderate block (MB) group
Drug: Rocuronium (DB group) — Post-tetanic count: 1-2 Titration of rocuronium dose
  Arms: Deep block (DB) group

SUMMARY:
The purpose of this study is to evaluated whether the depth of neuromuscular block may affect the unicon value of anesthetic depth monitoring system (ADMS).

ELIGIBILITY:
Inclusion Criteria:

* Gall bladder disease
* American Society of Anesthesiologist physical status 1 or 2

Exclusion Criteria:

* Pregnancy
* Body mass index < 16
* Body mass index >30
* Neuromuscular disease
* Previous intraabdominal surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Total infused dose of propofol | At 1 min after the anesthesia is finished

SECONDARY OUTCOMES:
Electromyographic index presented on the anesthetic depth monitoring system | Through study completion, an average of 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Seok Na, Principal Investigator — 82, Gumi 173
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea